CLINICAL TRIAL: NCT07247240
Title: Efficacy of Inhaled Nitric Oxide in Congenital Diaphragmatic Hernia With Early Pulmonary Hypertension
Brief Title: Efficacy of Inhaled Nitric Oxide in Congenital Diaphragmatic Hernia
Acronym: INOCDH
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Seoul National University Hospital (Other); Severance Hospital (Other); Chungnam National University Hospital (Other)
Responsible Party: Principal Investigator, Byong Sop Lee, Professor, Department of Pediatrics, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INOCDH_2025
Record Dates: First submitted 2025-09-30; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Congenital Diaphragmatic Hernia; Pulmonary Hypertension
Keywords: Congenital Diaphragmatic Hernia; Nitric Oxide; Pulmonary Hypertension
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital; Hypertension, Pulmonary | interventions — Inosine; Endothelium-Dependent Relaxing Factors

STUDY DESIGN:
Intervention Model Description: Assessment of Clinical Response After Administration of Inhaled Nitric Oxide in cases of CDH with Early Pulmonary Hypertension
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inhaled Nitric Oxide (Experimental): Administration of inhaled NO in newborn infants with CDH approaching predefined criteria of pulmonary hypertension and hypoxic respiratory failure
  Interventions: Drug: Inhaled Nitric Oxide

INTERVENTIONS:
Drug: Inhaled Nitric Oxide — Inhalation of nitric oxide for 30 minutes in CDH approaching predefined criteria of moderate to severe pulmonary hypertension and define the short-term response
  Other Names: iNO, Nitric Oxide gas

SUMMARY:
This multicenter, prospective, single-arm study aims to evaluate the efficacy of inhaled nitric oxide (iNO) in neonates with congenital diaphragmatic hernia (CDH) and early pulmonary hypertension. Short-term treatment response will be assessed by the changes in oxygenation index and other parameters including echocardiographic parameters at predefined intervals.

DETAILED DESCRIPTION:
Congenital diaphragmatic hernia (CDH) is a life-threatening congenital anomaly characterized by pulmonary hypoplasia and persistent pulmonary hypertension of the newborn (PPHN). Despite advances in neonatal intensive care, management of pulmonary hypertension remains a major challenge, and the role of inhaled nitric oxide (iNO) in this population is still controversial.

This study evaluates the therapeutic efficacy and physiological responses to iNO in late preterm (34 weeks of gestational age or more) or term neonates with Bochdalek-type CDH and severe pulmonary hypertension who require mechanical ventilation but are not placed on ECMO within 14 days of life.

iNO will be initiated at 20 ppm, and serial measurements of oxygenation index, arterial blood gas, vital signs, cerebral oxygen saturation (NIRS), and echocardiographic indices will be performed to evaluate the short-term treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Bochdalek type congenital diaphragmatic hernia
* Gestational age at 34 weeks or more and within 14 days after birth
* Hypoxic respiratory failure and pulmonary hypertension

Exclusion Criteria:

* Combined congenital heart disease requiring neonatal intervention or surgery
* Previous treatment of pulmonary vasodilators including inhaled nitric oxide
* on ECMO treatment

Ages: 1 Minute to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Response to inhaled nitric oxide | At 30-60 minutes after administration of inhaled nitric oxide.
  Participants were categorized as responders if their oxygenation index or FiO2 improved by more than 20% from baseline after administration of inhaled nitric oxide for at least 30 minutes.

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - Asan Medical Center, Seoul, Seoul
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Children's Hospital, Seoul
  - Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided